CLINICAL TRIAL: NCT03683888
Title: Effect of a Personalized Nutritional and Exercise Algorithm to Epicardial Fat in Patients With Obesity and Pre-Diabetes
Brief Title: Healthsnap on Epicardial Adipose Tissue Study
Acronym: HEATS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Gianluca Iacobellis, Professor of Medicine, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20171094
Record Dates: First submitted 2018-09-21; First posted 2018-09-25 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Obesity; Pre Diabetes
Keywords: epicardial fat
MeSH Terms: conditions — Obesity; Glucose Intolerance | interventions — Nutrition Assessment

STUDY DESIGN:
Intervention Model Description: Open-label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthsnap (Experimental): 50 patients will receive HealthSnap assessment in addition to their current treatment regardless of their participation into the study
  Interventions: Behavioral: HealthSnap
- Diet (Active Comparator): 50 patients will receive standard of care dietary counselling in addition to their current treatment regardless of their participation into the study
  Interventions: Behavioral: dietary counseling

INTERVENTIONS:
Behavioral: HealthSnap — HealthSnap provides personalized lifestyle reports and track progress over time using an electronic lifestyle record (ELR). HealthSnap Assessment is a simple, quick and not invasive tool that uses an algorithm that includes a questionnaire, physical measurements, dietary data and body fat indices
  Arms: Healthsnap
Behavioral: dietary counseling — Dietary counseling by RD. Low Calorie and/or Low Carb dietary plans will be discussed and provided to the study participant
  Arms: Diet

SUMMARY:
The purpose of this research study is to learn about the effectiveness of HealthSnap assessment, to reduce epicardial fat thickness. Excessive epicardial fat is associated with higher risk of developing diabetes and heart diseases. HealthSnap Assessment is a simple, quick and not invasive tool that will provide the patient with a personalized information nutritional and exercise plan.The use of HealthSnap in the clinical practice has not been evaluated, yet.

DETAILED DESCRIPTION:
This study will evaluate the practicality of adding the HealthSnap algorithm to the standard care of patients with overweight/obesity and pre-diabetes.

Participants will be recruited among the outpatient population who routinely refer to the Lennar Foundation Comprehensive Diabetes Center Outpatient Clinics, Division of Endocrinology, Diabetes and Metabolism University of Miami, for standard care and management of diabetes, obesity, overweight, hypertension, dyslipidemia.

Once patient eligibility and written consent are obtained, participant is then scheduled for the clinic visit through the University of Miami UChart (Epic) electronic system. The visits will be coordinated by the research coordinator. At each visit each patient will undergo:

* Full physical examination, body weight, height, waist and hip circumference, blood pressure (standard of care)
* Fasting blood glucose and haemoglobinA1c (HbA1c), lipid panel, comprehensive metabolic panel, fasting insulin, C-peptide and pro-insulin (all procedures are standard of care)
* Ultrasound assesment of epicardial fat, performed on site
* HealthSnap assessment performed on site (if randomized to the group receiving additional Healthnap)
* Standard of care dietary counselling performed on site by a registered dietitian (if randomized to the control group)

Study patients and controls will be contacted by the dietitian and/or HealthSnap supervisor once a week via telephone, or email (Uchart) or via online session (collaborate Ultra) to monitor their compliance and adherence to the exercise and dietary program.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) ≥ 27 kg/m2
* HbA1c 5.7-6.5% within 3 months the initial visit and/or
* Fasting blood glucose (FBG) 100-125 mg/dl within 3 months the initial visit and/or
* Family history for diabetes or CAD or dyslipidemia

Exclusion Criteria:

* • Type 1 diabetes

  * Pregnancy
  * Mental illness preventing correct use of HealthSnap
  * Physical inability to follow HealthSnap recommendations
  * Active infective and neoplastic diseases
  * No current diabetes medications with the exception of Metformin
  * Chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2020-09-10 (Actual); Study Completion 2020-09-10 (Actual)

PRIMARY OUTCOMES:
Epicardial fat thickness (EAT) | 3 months
  Change in ultrasound measured EAT

SECONDARY OUTCOMES:
Body Mass Index (BMI) | 3 months
  Change in BMI
Hemoglobin A1c (HbA1c) percentage (%) | 3 months
  Change in the HbA1c %

CONTACTS AND LOCATIONS:
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided